CLINICAL TRIAL: NCT04925830
Title: Inhibitory Training in Older Adults: a Biofeedback Study
Brief Title: Exploring the Impact of Biofeedback on the Inhibitory Control of Healthy Older Adults
Acronym: I-BF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Matthias Kliegel, Director, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 34_DT_Biofeedback
Record Dates: First submitted 2021-06-04; First posted 2021-06-14 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Inhibition
MeSH Terms: conditions — Inhibition, Psychological

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BF Group (Experimental): Participants of the BF group are connected with a plethysmograph and a respiration belt in order to assess HRV indices. HRV-BF is principally given by means of a vertical bar graph dynamically varying in height and two graphic curves referring to the heart rate (in beats per minute) and physiological breathing pattern, (inspiration and expiration). Each nirHEG- BF session occurs after a ten-minute pause from the end of the HRV-BF training. nirHEG-BF is principally given by means of a vertical bar graph dynamically varying in height and represented on a computer monitor. The height of the change according to the hemodynamic response measured at each of the three prefrontal points (Fp1, Fpz, Fp2) To maintain motivation, the bar graph is associated with a game-like animation (puzzle) signaling successful regulation, e.g. by forwarding motion of the pieces of a puzzle.
  Interventions: Behavioral: Heart rate variability biofeedback; haemoncephalography biofeedback
- No BF Group (No Intervention): The no BF group receive the same sensors and is exposed to the same environment of the BF group but real time biofeedback of physiological parameters (HRV and hemodynamic response) is deactivated so that participants can watch documentary videos without interruption.

INTERVENTIONS:
Behavioral: Heart rate variability biofeedback; haemoncephalography biofeedback — Ten 25-minute weekly heart rate variability biofeedback and 30 minute haemoencephalogrphy biofeedback sessions
  Arms: BF Group

SUMMARY:
Inhibitory control refers to the conscious and voluntary suppression of predominant responses when they are automatic, inappropriate, or incorrect. Inhibitory control plays a key role in self-regulation and self-control behaviors in many different areas of everyday life. During aging, their decline would impact executive functioning and mental health.

Recently, physiological training methods including heart rate variability biofeedback (HRV-BF), based on heart rate and respiration measurements, and hemoencephalography biofeedback (nirHEG NF), based on the hemodynamic response of some prefrontal regions, have proven to have a positive impact on executive functions. In this study, subjects of the experimental group were exposed to biofeedback training during 10 sessions, once a week, and their results compared to those of the control group, which did not receive biofeedback training.

This study aims to explore the impact of training that combines two innovative techniques, such as heart rate variability biofeedback and hemoencephalography biofeedback on the inhibitory control of older adults. We expect positive effects of biofeedback training on the inhibition tasks and the targeted physiological parameters.

Primary objective - We intend to demonstrate that heart rate variability biofeedback training coupled with hemoencephalography biofeedback training can be effective methods to counteract the decline of inhibitory control in older adults.

Secondary objective - We intend to demonstrate that heart rate variability biofeedback and hemoencephalography biofeedback can effectively increase heart rate variability and blood flood oxygenation.

DETAILED DESCRIPTION:
This is a pilot, randomized controlled study that aims to explore the effects of the combination of two interventions, HRV-BF and nirHEG neurofeedback, on the inhibitory control of healthy older adults. The study is thus designed with two parallel groups: the experimental group will receive sessions of HRV-BF and nirHEG NF whereas the control group will receive sessions in which visual biofeedback will be disabled.

The three tasks used in the present study to appraise inhibitory control are Go/no Go, The Arrow task and Stroop task whereas impulsive behaviour will be evaluated with the UPPS scale. In addition, the feeling of self-efficacity and the attitude toward stereotypes will also be assessed with respectively the Self-efficacity scale and l'Echelle du moral. All these tasks will be administered at pretest and posttest intervention.

Procedures Healthy older adults will be recruited by public advertisements and flyers posted at the Universities of Geneva, in sport clubs and various seniors associations.

After a verbal consent and an initial telephone interview (anamnestic questionnaire and F-TICS-m-Telephone Interview for Cognitive Status questionnaire, Vercambre et al.,2010), the eligible participants will be asked to attend a first visit during which written informed consent will be obtained.

After confirmation of eligibility and enrolment, the 50 selected participants will be randomly assigned to an experimental or a control group each group counting about 25 subjects. First, both study groups will be evaluated with a battery of inhibition and psychological testing. Then, the experimental group (n=25) will receive 10 biofeedback training sessions (heart rate variability plus hemoencephalography neurofeedback, 1 hour session, once a week for 10 weeks. The control group (n=25) will receive sessions in which visual biofeedback will be disabled.

Both study groups will be evaluated at 2 points - pre and post training on inhibitory control, impulsivity, heart rate variability levels, hemodynamic response, feeling of self-efficacity and attitude toward aging.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* 65 to 80 years old
* Native French speakers or speaking French for over 5 years

Exclusion Criteria:

* Adults who report <27 on TICS (Telephone Interview for Cognitive Status questionnaire)
* Adults that report a history of major neurological or psychiatric illness in the present or the past
* Use of psychotropic drugs

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2021-06-17 (Actual); Study Completion 2021-06-17 (Actual)

PRIMARY OUTCOMES:
Change in interference score (milliseconds) | Pre-intervention (week 1) - Post-intervention (week 13)
  Between group post-pre interference score change (reaction time) in Arrow task
Change in inhibitory response (milliseconds) | Pre-intervention (week 1) - Post-intervention (week 13)
  Between group post-pre reaction time change in GO no GO
Change in interference score (seconds) | Pre-test (week 1) - Posttest (week 13)
  Between group post-pre interference score in Stroop task

SECONDARY OUTCOMES:
Heart rate variability changes | HRV-baseline (week 2) - HRV-posttest (week 13)
  Between group post-pre change in heart rate variability values (RMSSD, LF, HF)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Kliegel, Professor, Principal Investigator — University of Geneva
Locations (1):
- Center for the Interdisciplinary Study of Gerontology and Vulnerabilities (CIGEV), Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No